CLINICAL TRIAL: NCT04519229
Title: Child-Parent Psychotherapy for Children 0-6 Years Old With Experiences of Adverse Life Events - a Feasibility Study for Children in Foster Care
Brief Title: Child-Parent Psychotherapy - a Feasibility Study for Children in Foster Care
Status: Enrolling by invitation | Type: Observational
Sponsor: Kronoberg County Council (Other Government)
Collaborators: Stiftelsen Allmänna Barnhuset (Unknown)
Responsible Party: Sponsor
Other Study IDs: RK/30062020
Record Dates: First submitted 2020-07-09; First posted 2020-08-19 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Child Abuse; Child Neglect; Post-Traumatic Stress Disorder in Children; Parent-Child Relations
Keywords: Children; Adverse childhood events; Post traumatic stress; Children in foster care; Psychotherapy

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children in fostercare in CPP-treatment: Children in foster care taking part in Child-Parent Psychotherapy
  Interventions: Behavioral: Child-Parent Psychotherapy

INTERVENTIONS:
Behavioral: Child-Parent Psychotherapy — Relationship-based trauma focused psychotherapy for Children 0-6 years old and their caregivers. The objective is to decrease symptoms of post-traumatic tress and re-establish a secure attachment for the child and good caregiving from the caregiver/s.

SUMMARY:
Children in foster care have an increased risk of exposure to adverse experiences during childhood and across the lifespan. In current studies of interventions children in foster care are often excluded, or they are too few to be included in statistical analyses of outcomes. As a consequence, knowledge on feasibility of treatment methods for some of the most exposed and maltreated children in society is sparse.

Child-Parent Psychotherapy (CPP) is an intervention for children 0-6 years who have been exposed to adverse and traumatic events. CPP is currently being implemented in Sweden. The aim of this study is to investigate the feasibility of CPP for children in foster care.

DETAILED DESCRIPTION:
Aim. The aim of the current study is to investigate the feasibility of CPP for young children who have an increased risk of exposure to adverse and traumatic experiences with negative effects on their health and development. Feasibility will be conceptualized as acceptance of the method by therapists, caregivers, and children; practical applications of the method; any need for modifications; and observed outcomes.

Research questions The main research question is: Is CPP feasible for children in foster care? Additional research questions are: 1) How do children in foster care experience participating in CPP? 2) How do foster parents experience participating in CPP? 3) How do clinicians experience using CPP with children in foster care and their caregivers? 4) What outcomes can be observed in treatment with children in foster care in terms of increased psychological health in children and foster parents; decrease in symptoms of post-traumatic stress in children and foster parents; and foster parents' experiences of their caregiving capacity and relationship with the child.

Method Design. The project has a naturalistic mixed-methods study design. Qualitative and quantitative research methods will be used to collect and analyze data. Qualitative data concerning childrens', caregivers', and clinicians' experiences of the treatment method as well as quantitative data concerning practical applications of the method, any modifications made, and reported levels of symptoms will be studied.

Participants. Nine agencies in different regions of Sweden offering CPP as part of their regular services have accepted to participate in the study. Participants are consecutively recruited at the participating agencies. Inclusion will be terminated when 20 children have been included (whereof at least 12 children aged 3-6 years).

Procedure. At treatment start caregivers and custodians (this can include foster parents, social services, and biological parents) will be informed about the study and asked for consent to participate. Because of their low age children aged 3-6 will be informed and asked for consent to participate in connection to the interviews. Quantitative data will be collected by self-report instruments completed by the foster parents before treatment and after 20 sessions or at termination, if treatment if terminated earlier. Participation, fidelity, and modifications are registered by clinicians continuously. Foster parents and clinicians will be asked to schedule interviews by one of the researchers in the project after 20 sessions or at termination, if treatment if terminated earlier.

Background information. Demographical and background data will be collected using a form designed for this purpose, before treatment and after 20 sessions or at termination, if treatment is terminated earlier.

Instrument. Qualitative interviews focusing acceptance and experiences of the method will be conducted with children, foster parents, and clinicians. The interviews will be conducted by child psychologists experienced in clinical treatment as well as in research with families with young children in in difficult life situations. The interviews will be recorded and transcribed verbatim. Clinicians will register participation, fidelity, and any modifications after each treatment session in a log-book. Quantitative data on outcome concerning exposure, symptoms of post-traumatic stress, psychological health, and caregiving experiences will be collected by self-report instruments completed by foster parents before treatment and after 20 sessions or at termination, if treatment is terminated earlier.

Analyses. The interviews will be analyzed by thematic analysis or interpretative phenomenological analysis, according to the applicability in relation to the research questions and data collected. Descriptive statistical methods will be used to describe exposure, symptoms pre- and post-treatment, and treatment modifications made. Non-parametric statistical methods will be used to analyze and describe indications concerning outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age 0-6 years
* being offered Child-Parent Psychotherapy as part of their regular treatment

Exclusion Criteria:

* Families in need of translator for interviews.

Ages: 0 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children in foster care offered Child-Parent Psychotherapy at any of the nine participating agencies.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-06-30 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline score on the Strengths and Difficulties Questionnaire - Parent version at 20 completed sessions or at termination of intervention if terminated earlier. | After 20 completed sessions or immediately after termination of the intervention, if terminated earlier than 20 sessions
  Caregiver report of child psychopathology. Minimum score 0, maximum score 40, higher score indicating worse outcome.
Change from baseline score on the Trauma Symptom Checklist for Young Children at 20 completed sessions or at termination of intervention if terminated earlier. | After 20 completed sessions or immediately after termination of the intervention, if terminated earlier than 20 sessions
  Caregiver report of child symptoms of post-traumatic stress. Minimum score 90, maximum score 360, higher score indicating worse outcome.
Change from baseline score on the Linköping Youth Life Experiences Scale at 20 completed sessions or at termination of intervention if terminated earlier. | After 20 completed sessions or immediately after termination of the intervention, if terminated earlier than 20 sessions
  Caregiver report of child exposure to traumatic and adverse life events. Minimum score 0, maximum score 41, higher score indicating worse outcome.
Change from baseline score on the Child-Parent Psychotherapy Symptom Screener at 20 completed sessions or at termination of intervention if terminated earlier. | After 20 completed sessions or immediately after termination of the intervention, if terminated earlier than 20 sessions
  Caregiver report of child symptoms of post-traumatic reactions. Minimum score 0, maximum score 93, higher score indicating worse outcome.

SECONDARY OUTCOMES:
Change from baseline score on the Hopkins Symptom Check List-25 at 20 completed sessions or at termination of intervention if terminated earlier. | After 20 completed sessions or immediately after termination of the intervention, if terminated earlier than 20 sessions
  Caregiver report of psychological distress and symptoms. Minimum score 0, maximum score 100, higher score indicating worse outcome.
Change from baseline score on the Impact of Event Scale-Revised at 20 completed sessions or at termination of intervention if terminated earlier. | After 20 completed sessions or immediately after termination of the intervention, if terminated earlier than 20 sessions
  Caregiver report of symptoms of post-traumatic stress. Minimum score 0, maximum score 80, higher score indicating worse outcome.
Change from baseline score on the Life Incidence of Traumatic Events Questionnaire at 20 completed sessions or at termination of intervention if terminated earlier. | After 20 completed sessions or immediately after termination of the intervention, if terminated earlier than 20 sessions
  Caregiver report of exposure to traumatic and adverse life events. Minimum score 0, maximum score 41, higher score indicating worse outcome.
Change from baseline score on the Caregiving Helplessness Questionnaire at 20 completed sessions or at termination of intervention if terminated earlier. | After 20 completed sessions or immediately after termination of the intervention, if terminated earlier than 20 sessions
  Caregiver report on caregiving experiences. Minimum score 18, maximum score 90, higher score indicating worse outcome.

OTHER OUTCOMES:
Adherence | After 20 completed sessions or immediately after termination of the intervention if terminated earlier than 20 sessions
  Log of clinicians' ratings of fidelity to the method of Child-Parent Psychotherapy and adaptions immediately after each session, up to 20 times
Childrens' experiences of participating in Child-Parent Psychotherapy | After 20 completed sessions or immediately after termination of the intervention if terminated earlier than 20 sessions
  Qualitative data from interviews with children 3-6 years old
Foster parents' experiences of participating in Child-Parent Psychotherapy | After 20 completed sessions or immediately after termination of the intervention if terminated earlier than 20 sessions
  Qualitative data from interviews with foster parents
Clinicians' experiences of working with Child-Parent Psychotherapy with Children in foster care | After 20 completed sessions or immediately after termination of the intervention if terminated earlier than 20 sessions
  Qualitative data from interviews with clinicians

CONTACTS AND LOCATIONS:
Overall Officials: Karin Pernebo, PhD, Study Director — Department of Psychology, Linnaeus University, Sweden and Department of Research and Development, Region Kronoberg, Sweden
Locations (1):
- Department of Research and Development, Region Kronoberg, Vaxjo, Sweden

IPD SHARING:
Plan to Share IPD: No